CLINICAL TRIAL: NCT01752946
Title: A Registry Study of Shuxuening (a Chinese Medicine Injection) Used in Hospitals in China
Brief Title: A Registry Study of Shuxuening Injection Used in Hospitals in China
Acronym: RSCMI-VII
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: China Academy of Chinese Medical Sciences (Other)
Collaborators: Beijing University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, Xie Yanming, Deputy Director, China Academy of Chinese Medical Sciences
Other Study IDs: 2009zx09502-030-07
Record Dates: First submitted 2012-12-15; First posted 2012-12-19 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2012-12

CONDITIONS: Coronary Disease; Intracranial Embolism; Stroke; Angina Pectoris; Vasospasm
MeSH Terms: conditions — Coronary Disease; Intracranial Embolism; Stroke; Angina Pectoris

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is get to know what and how Shuxuening injection in hospital results in adverse events or adverse drug reactions from a cohort event monitoring.

DETAILED DESCRIPTION:
Ginkgo leaf is major component of Shuxuening injection. Although some western countries product similar injections and use them, Shuxuening injection also regarded as Chinese medicine injection. As a TCM injection, the most important thing is how to safety use it in practice.

In order to improving monitoring adverse events or adverse drug reaction of Chinese medicine injection in hospital, registry study is suitable method in this area. Otherwise, nested case control study is used to find out the mechanism of allergic reaction.

Calculate the incidence of adverse events or adverse drug reaction is one of the main aims for this study. Safety surveillance on Chinese Medicine injection is an important problem that needs to be sorted out through large sample observational study.

According to the 'rule of three', 30,000 cases need to be registered at least. The aim population is who using Shuxuening injection's during inpatient time from December 2012 to December 2014.

Data will be collected for three departments as following:

Form A (green): demographic information ；Form B (pink): adverse drug events/reaction； Form C (white): extracted information from hospital information system and laboratory information system.

ELIGIBILITY:
Inclusion Criteria:

* Patients using Shuxuening injection from 2012 to 2014

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: According to the 'rule of three', 30,000 cases need to be registered at least. The aim population is who using Shuxuening injection's during inpatient time from December 2012 to December.2014 in more than 30 hospitals in China.
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2012-10; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Shuxuening injection's ADRs and factors contributed to the occurrence of the adverse reaction | to assess Shuxuening's "adverse event" and "drug adverse reaction" during patients' hospital stay, administration information of Shuxuening will be registered every day. The registry procedure will last 2 years only for patients using Shuxuening.
  All participants will be followed for the duration of hospital stay, an expected average of 2 weeks. Patients using Shuxuening will be registered on a registration form including disease background, Shuxuening's administration, and extraction information from hospital information system. When the patients occurs allergic reaction during using Shuxuening injection, it also need to collect patient's biological samples. An adverse event or drug adverse reaction form also will be used to describe any doubted symptoms or signs from patients. A judgment will be made by doctors directly and a further analysis will be conducted by researchers to decide those potential side-effects of Shuxuening injection.

CONTACTS AND LOCATIONS:
Overall Officials: Yan M Xie, BA, Principal Investigator — Institute of Basic Research in Clinical Medicine, China Academy of Chinese Medical Sciences